CLINICAL TRIAL: NCT00403299
Title: Multidetector Computer Tomography of the Coronary Arteries in Heart Transplanted Patients
Brief Title: MDCT of the Coronary Arteries in Heart Transplanted Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: S-05203
Record Dates: First submitted 2006-11-22; First posted 2006-11-23 (Estimated); Last update posted 2011-07-06 (Estimated); Status verified 2008-04

CONDITIONS: Coronary Artery Disease
Keywords: Coronary artery disease; Cardiac transplantation; Coronary artery disease in heart transplanted patients
MeSH Terms: conditions — Coronary Artery Disease

INTERVENTIONS:
Procedure: MDCT of the coronary arteries.

SUMMARY:
Heart transplanted patients often develop coronary artery disease and therefore have their coronary arteries examined with coronary angiography once a year.The purpose of the study is to validate computer tomography of the coronary arteries against coronary angiography and intravascular ultrasound in heart transplanted patients. Additionally the association between different inflammatory markers and the development of CAD specific to heart transplanted patients will be studied.

DETAILED DESCRIPTION:
Heart transplanted patients (HTx) often develop coronary artery disease (CAD) which is a major cause of graft failure and death in this group of patients. Therefore, heart transplanted patients have their coronary arteries examined annually. At present this is being done with coronary angiography. Recent development of the computed tomography (CT) technology has made it possible to examine the coronary arteries with CT angiography (CTA), which is a non-invasive method. The goal of the study is to validate CTA against coronary angiography.

Coronary artery disease lesions in heart transplanted patients differ from CAD lesions in native hearts. HTx patients develop diffuse intimal thickening affecting the whole length of the vessel starting in the periphery. These lesions specific to HTx patients are not depicted on coronary angiography. The second aim of this study is to compare the accuracy of CTA depicting such lesions with the gold-standard, intravascular ultrasound.

The third aim of this study is to study the association between different inflammatory markers and the development of CAD specific to heart transplanted patients.

ELIGIBILITY:
Inclusion Criteria:

* Heart transplanted patient
* Age 18 or above.

Exclusion Criteria:

* Heart transplantation less than a year ago.
* Renal insufficiency with estimated creatinine clearance < 50 ml/min.
* History of contrast induced nephropathy.
* Known allergic reaction to CT contrast.
* Pregnancy
* Atrial Fibrillation
* Severe heart failure NYHA class IV.
* Hypotension (systolic blood pressure (BP) < 100 mmHg and/or diastolic BP<50 mmHg) or hemodynamic unstable patients.
* Severe pulmonary disease making the patient unable to hold his/her breath in more than 10 seconds.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2006-03; Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Coronary artery disease found on computer tomography examination at the date of examination.

SECONDARY OUTCOMES:
Coronary artery disease found on coronary angiography at the date of examination.
Coronary artery disease found on intravascular ultrasound examination at the date of examination.

CONTACTS AND LOCATIONS:
Overall Officials: Anne Günther, MD, Principal Investigator — Oslo University Hospital
Locations (1):
- Rikshospitalet-Radiumhospitalet HF, Oslo, Norway